CLINICAL TRIAL: NCT06892600
Title: Combined General and Spinal Anesthesia Compared to General Anesthesia During Laparoscopic Surgery : a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Pryambodho Pryambodho, MD, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23060823
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Laparoscopic Abdominal Surgery; Spinal Anesthesia; General Anesthesia Using Endotracheal Intubation
Keywords: laparoscopy; combined spinal and general anesthesia; abdominal laparoscopic surgery; opioid consumption; spinal anesthesia
MeSH Terms: interventions — Anesthesia, General; Control Groups

STUDY DESIGN:
Intervention Model Description: Two parallel groups - intervention and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined group (Experimental): Combined spinal anesthesia and general anesthesia Spinal anesthesia is given at L2-3/L3-4 level with Quincke 27G spinal needle, with 10 mg of Bupivacaine heavy 0.5% General anesthesia is induced with lidocaine 1.5mg/kg, fentanyl 2 mcg/kg, propofol 2 mg/kg, rocuronium 0.6 mg/kg
  Interventions: Drug: Combined Spinal anesthesia (heavy bupivacaine 0.5%) and General anesthesia
- Control (Active Comparator): General anesthesia only Lidocaine 1.5mg/kg, fentanyl 2 mcg/kg, propofol 2 mg/kg, rocuronium 0.6 mg/kg
  Interventions: Drug: General Anesthesia (control group)

INTERVENTIONS:
Drug: Combined Spinal anesthesia (heavy bupivacaine 0.5%) and General anesthesia — Combined spinal and general anesthesia Spinal anesthesia with Bupivacaine heavy 0.5% 10 mg General anesthesia with Lidocaine 1.5mg/kg, Fentanyl 2 mcg/kg, propofol 2 mg/kg, Rocuronium 0.6 mg/kg
  Arms: Combined group
Drug: General Anesthesia (control group) — Lidocaine 1.5mg/kg, fentanyl 2 mcg/kg, propofol 2 mg/kg, rocuronium 0,6 mg/kg
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if combining spinal and general anesthesia is better than general anesthesia alone for abdominal laparoscopic surgery in adults. The main questions it aims to answer are:

Does combining spinal and general anesthesia provide better stability compared to general anesthesia alone during abdominal laparoscopic surgery? Does combining spinal and general anesthesia lead to less opioid consumption compared to general anesthesia alone for abdominal laparoscopic surgery?

Participants will:

Be randomized and allocated to either spinal and general anesthesia (combined) group vs general anesthesia (control) group In the combined group, participants will be given a spinal anesthesia followed by general anesthesia, compared to general anesthesia alone in the control group.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) 1-2
* BMI ≤ 30 kg/m2
* Adults (18-64 years old) who will undergo elective abdominal laparoscopic surgery (digestive surgery, gynecologic surgery or urologic surgery)
* Willing to participate in this study

Exclusion Criteria:

* Cardiovascular disease (uncontrolled stage 2 hypertension, AV block, valvular heart disease, heart failure or arrythmia)
* Cerebrovascular disease (within < 3 months)
* Infection at the proposed site of spinal injection
* Coagulopathy
* Elevated intracranial pressure
* Severe kidney or liver dysfunction

Drop out criteria:

* Anesthesia duration > 6 hours
* Intraoperative emergency
* Conversion to open laparotomy
* Spinal complications (shock, anaphylaxis, seizure or high spinal)
* Failed spinal (2 attempts)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Throughout the surgery
  Fentanyl dosage in mcg used during the procedure
Post-operative pain score | Within 24 hours after surgery
  Post operative pain score
Hemodynamic stability | During the surgery
  Mean arterial pressure (MAP) after insufflation variation of < 20% compared to MAP after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Pryambodho Pryambodho, MD, Anesthesiologist, Principal Investigator — Indonesia University
Locations (1):
- Cipto mangunkusumo general hospital, Jakarta, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No
The data may be available upon request if needed.